CLINICAL TRIAL: NCT01453257
Title: A Phase 2 Study of Target-Guided Personalized Chemotherapy in Metastatic Colorectal Cancer Patients
Brief Title: Study of Target-Guided Chemotherapy in Metastatic Colorectal Patients
Acronym: TT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Hospital de Madrid (Other)
Responsible Party: Principal Investigator, Sofia Perea, PharmD, PhD, Fundación Hospital de mADRID, Grupo Hospital de Madrid
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C62 202-878
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Progression Free Survival
Keywords: Molecular Targets; Personalize Treatment; Colon Cancer; Complete Response Rate
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy treatment (Experimental): Tailored chemotherapy by Therapeutic Targets
  Interventions: Drug: Tailored Chemotherapy

INTERVENTIONS:
Drug: Tailored Chemotherapy — Patients will be treated with Folfox, Folfiri, Xelox or Xeliri and Cetuximab or Bevacizumab at usual doses tailored by:
  K-ras native: Cetuximab. K-ras mutated: Bevacizumab Topoisomera 1 positive ( Topo-1): Irinotecan Topo-1 positive and ERCC-1 negative: oxaliplatin Topo-1 1 negative and ERCC-1 positive: investigator option Thimidylate synthase (TS) positive: No Fluoropyrimidines (FLP) TS negative: FLP Thimidylate phosphorylasa (TP) positive: Capecitabine TP negative: 5-FU
  Other Names: Biomarker selection; Therapeutic Targets chemotherapy

SUMMARY:
Treatment options for patients with colorectal cancer (CRC) have increased in the last years. However, there are no validated prospective molecular markers in CRC to select which agents are better to treat any individual case. The conventional first-line treatment in CRC patients in clinical studies get a proportion of patients free of progression at 12 months ranging from 35-40% with a median of 9 months of free disease progression.

The aim of this study is to demonstrate that the identification of therapeutic targets in real time and their prospectively use to customize the treatment get a proportion of colorectal metastatic patients patients free of progression disease at 12 months of 50%.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal adenocarcinoma stage IV patients.
* ECOG= 0-1
* Age > 18 years.
* Fit to receive chemotherapy treatment
* Availability of tumor tissue or possibility of a tumor biopsy to determine therapeutic targets.
* Adequate renal (Cr < 1,5 mg/d), liver (bilirubin≤1,5 mg/dl, AST and ALT ≤ 3.0 x the upper limit of normal) and normal bone marrow function ( absolute neutrophil count ≥ 1500/µl, hemoglobin ≥ 9.0g/dl and a platelet count of ≥ 100.000/µl)

Exclusion Criteria:

* Contraindication for the administration of any of the drugs used in the study including capecitabine, irinotecan, oxaliplatin, cetuximab or bevacizumab.
* Previous Chemotherapy treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
PFS | 12 months

SECONDARY OUTCOMES:
Complete Response Rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cubillo, Md PhD, Principal Investigator — Grupo Hospital madrid
Locations (1):
- Centro Integral Oncológico Clara campal, Madrid, Madrid, Spain